CLINICAL TRIAL: NCT01965938
Title: RIFL (Rigid and Flexing Laryngoscope) vs. Fiberoptic Bronchoscope: A Comparison of the Ease of Use During Intubation on Difficult Airways
Brief Title: RIFL (Rigid and Flexing Laryngoscope) vs. Fiberoptic Bronchoscope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Bret Alvis, Clinical Fellow, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 121408
Record Dates: First submitted 2013-10-16; First posted 2013-10-18 (Estimated); Results first posted 2017-01-05 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2016-10

CONDITIONS: Intubation; Difficult

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RIFL (Rigid and Flexing Laryngoscope) (Active Comparator): Patients in the RIFL group will undergo bronchoscopy using the Rigid and Flexing Laryngoscope. Once the carina is visualized with the bronchoscope, the endotracheal tube will be advanced, and the bronchoscope removed.
  Interventions: Device: RIFL (Rigid and Flexing Laryngoscope)
- Fiberoptic Bronchoscope (Other): Patients in the control group will undergo bronchoscopy using the flexible fiberoptic bronchoscope. Once the carina is visualized with the bronchoscope, the endotracheal tube will be advanced, and the bronchoscope removed.
  Interventions: Device: Fiberoptic Bronchoscope

INTERVENTIONS:
Device: RIFL (Rigid and Flexing Laryngoscope) — Patients in the RIFL group will undergo bronchoscopy using the Rigid and Flexing Laryngoscope. Once the carina is visualized with the bronchoscope, the endotracheal tube will be advanced, and the bronchoscope removed.
  Other Names: Video RIFL RIgid Flexible Laryngoscope; AI Medical Devices, Inc
  Arms: RIFL (Rigid and Flexing Laryngoscope)
Device: Fiberoptic Bronchoscope — Patients in the control group will undergo bronchoscopy using the flexible fiberoptic bronchoscope. Once the carina is visualized with the bronchoscope, the endotracheal tube will be advanced, and the bronchoscope removed.
  Arms: Fiberoptic Bronchoscope

SUMMARY:
We will conduct a randomized trial comparing the success rate and time to intubation using the RIFL vs. the fiberoptic bronchoscope, as the latter is commonly held to be the gold standard of difficult airway devices. Specifically, we wish to compare the of intubation between the two devices in patients with potentially difficult airways as defined by an oropharyngeal class 3-4, BMI greater than 35, or in patients with a history of difficult intubation using direct laryngoscopy.

DETAILED DESCRIPTION:
Patients who require general anesthesia with endotracheal intubation will be identified the night prior to their surgery based upon the examination documented in their preoperative history and physical. If their body mass index achieves a calculated score of 35 or greater or they have an oropharyngeal class 4 airway then they will qualify to participate.

After written informed consent is obtained, The intubation method would be randomized as one of two groups: intubation via use of the fiberoptic bronchoscope or the RIFL. The intubation attempt will be terminated if the SpO2 <90, HR<50, there is traumatic injury, or time > 100sec. If terminated, the patient will be mask ventilated and the attending anesthesiologist would determine the subsequent technique that will be used for airway management.

ELIGIBILITY:
Inclusion Criteria:

Patients with known or suspected difficult airways defined as:

* patients with an oropharyngeal score of 3 or 4
* patients whose body mass index calculates greater to or equal to 35

Exclusion Criteria:

* Patients who necessitate an awake fiberoptic intubation or a rapid sequence intubation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2012-09; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bret Alvis, M.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RIFL (Rigid and Flexing Laryngoscope) | Fiberoptic Bronchoscope
Started | 21 | 20
Completed | 20 | 20
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RIFL (Rigid and Flexing Laryngoscope) | Fiberoptic Bronchoscope | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (15) | 49 (12) | 49.5 (14)
Gender [Count of Participants; unit: Participants]
  Female | 10 | 13 | 23
  Male | 10 | 7 | 17
Mallampati Class (N) [Number; unit: participants] — Mallampati Class
  Class I: Soft palate, fauces, uvula, pillars visible Class II: Soft palate, fauces, uvula visible Class III: Soft palate, base of uvula visible Class IV: Soft palate not visible at all
  A high Mallampati score (class 3 or 4) is associated with more difficult intubation
  participants
    Class 1 | 3 | 1 | 4
    Class 2 | 2 | 3 | 5
    Class 3 | 6 | 7 | 13
    Class 4 | 9 | 9 | 18
Anticipated Difficult airway [Number; unit: participants] — Anticipated difficult airway was defined as patients who met one or more of the following criteria: past history of documented difficult intubation, Mallampati Score ≥3, and a body mass index (BMI)≥35.
  participants
    Yes | 9 | 6 | 15
    No | 11 | 14 | 25

OUTCOME MEASURES:

1. Primary Outcome: Time Until Proper Endotracheal Tube Placement
Description: Time (in seconds) from first placement of the intubating scope in the oral cavity until proper endotracheal tube placement is confirmed by the presence of End Tidal Co2 (etCO2). Time to successful intubation was defined as the period from when the tip of the RIFL or FOB passed the incisors until withdrawal past that same point after successful intubation.
Time Frame: usually <100 seconds
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | RIFL (Rigid and Flexing Laryngoscope) | Fiberoptic Bronchoscope
Number analyzed (Participants) | 20 | 20
seconds | 49 [24 to 73] | 64 [40 to 120]

2. Secondary Outcome: Number of Participants With Successful Intubation
Description: Successful intubation defined as confirming tube placement by the presence of etCO2;
Time Frame: <100 seconds
Measure: Number; unit: participants
Arm/Group | RIFL (Rigid and Flexing Laryngoscope) | Fiberoptic Bronchoscope
Number analyzed (Participants) | 20 | 20
participants | 20 | 20

3. Secondary Outcome: Number of Attempts Performed During Airway Management
Time Frame: <100 seconds
Measure: Mean (Standard Deviation); unit: number attempts
Arm/Group | RIFL (Rigid and Flexing Laryngoscope) | Fiberoptic Bronchoscope
Number analyzed (Participants) | 20 | 20
number attempts | 1.1 (0.3) | 1.2 (0.5)

4. Secondary Outcome: Grade of Glottic View
Description: According to McCormack and Lehane
Time Frame: <100 seconds
Population: data was not collected
Arm/Group | RIFL (Rigid and Flexing Laryngoscope) | Fiberoptic Bronchoscope
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Assistance Maneuvers, if Any, Provided by the Attending Anesthesiologist
Description: Number of patients that required Assistance Maneuvers provided by the attending anesthesiologist such as jaw lift, tongue protrusion, laryngeal pressure, etc
Time Frame: <100 seconds
Measure: Number; unit: participants
Arm/Group | RIFL (Rigid and Flexing Laryngoscope) | Fiberoptic Bronchoscope
Number analyzed (Participants) | 20 | 20
participants | 2 | 16

6. Secondary Outcome: Lowest Pulse Oximetry Saturation Value Reading During Intubation
Description: Lowest pulse oximetry saturation value reading collected from any participant during intubation
Time Frame: <100 seconds
Measure: Number; unit: percentage of saturated hemoglobin
Arm/Group | RIFL (Rigid and Flexing Laryngoscope) | Fiberoptic Bronchoscope
Number analyzed (Participants) | 20 | 20
percentage of saturated hemoglobin | 100 | 100

7. Other Pre Specified Outcome: Oropharyngeal Injuries
Description: Number of patients with any notation of any trauma to lips, teeth, soft tissue, etc.
Time Frame: 24 hours
Measure: Number; unit: participants
Arm/Group | RIFL (Rigid and Flexing Laryngoscope) | Fiberoptic Bronchoscope
Number analyzed (Participants) | 20 | 20
participants | 2 | 3

8. Secondary Outcome: Alternate Device Used
Time Frame: <100 seconds
Measure: Number; unit: number times an alternate device used
Arm/Group | RIFL (Rigid and Flexing Laryngoscope) | Fiberoptic Bronchoscope
Number analyzed (Participants) | 20 | 20
number times an alternate device used | 0 | 0

ADVERSE EVENTS:
Time Frame: During hospital stay (approximately 1-4 days)
Arm/Group | RIFL (Rigid and Flexing Laryngoscope) | Fiberoptic Bronchoscope
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 2/20 | 3/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RIFL (Rigid and Flexing Laryngoscope) (N=20) | Fiberoptic Bronchoscope (N=20)
Oropharyngeal injuries (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No